CLINICAL TRIAL: NCT03426839
Title: Haemostasis Management of Patients Undergoing Abdominal Aortic Procedures Associated With High Bleeding Risk
Brief Title: Haemostasis Management of Abdominal Aortic Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Upecs
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Abdominal Aortic Aneurism; Abdominal Aortic Rupture; Perioperative/Postoperative Complications; Surgical Blood Loss
Keywords: hemostatic techniques; perioperative hemorrhage; platelet function test; point of care technology; thromboelastometry; vascular surgical procedures
MeSH Terms: conditions — Postoperative Complications; Blood Loss, Surgical | interventions — Blood Coagulation Tests

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to each of two treatment groups using sealed envelopes:
  * Patient group 1: haemostasis strategy guided by conventional coagulation tests.
  * Patient group 2: transfusion algorithm guided by viscoelastic POC tests and algorithms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): In the conventional group (group 1) haemostasis strategy guided by conventional coagulation tests will be carried out.
  Interventions: Diagnostic Test: Coagulation tests
- Point of care group (Active Comparator): In the point of care group (group 2) transfusion algorithms guided by point-of-care (POC) tests will be applied. We will use viscoelastic thromboelastometry and impedance aggregometry.
  Interventions: Diagnostic Test: Coagulation tests

INTERVENTIONS:
Diagnostic Test: Coagulation tests
  Other Names: Conventional coagulation tests; Point of care coagulation tests

SUMMARY:
Comparative study on efficacy of haemostatic therapy guided either by standard laboratory coagulation parameters or point-of-care testing in patients undergoing vascular surgical procedures. We investigate the amount of perioperative bleeding and the number of blood product used.

Inclusion criteria Patients scheduled for elective and acute open aorta surgery or undergoing acute aorta surgery with minimally invasive techniques and were provided treatment in the operating theatre and/or ICU attached to perioperative care, they must be at least 18 years of age and written informed consent was obtained from the patient or his/her legal representative.

Randomisation technique Patients will be randomly assigned to each of two treatment groups using sealed envelopes. In group 1 (G1) haemostasis strategy guided by conventional coagulation tests, while in group 2 (G2) transfusion algorithms guided by point-of-care (POC) tests will be carried out.

Sampling techniques and measurements

For assessment of monitored parameters shall be used arterial or venous blood depending on the catheter placed preoperatively. In case of the above mentioned vascular surgical procedures, all patients will receive arterial cannula routinely, and, depending on the extension of procedure, as appropriate, a central venous catheter will be inserted as well. Sampling in the patient groups shall be performed as follows:

* pre- and postoperative evaluation of standard laboratory parameters in all patients
* evaluation of standard laboratory parameters and arterial Astrup test during and after surgery in group 1, if the blood loss volume reaches 1,5 ml/kg/minute during 20 minutes
* in case of elective surgery: thromboelastometry and arterial Astrup test during and after surgery in group 2 if the blood loss volume reaches 1,5 ml/kg/minute during 20 minutes
* in case of acute surgery: thromboelastometry and arterial Astrup test before, during and after surgery in group 2
* in case of positive anamnesis, preoperative platelet aggregation test in both groups Besides the above samplings, routine lab tests (blood gas, blood count, sodium (Na), potassium (K), parameters of renal and liver function, clotting and inflammation, lactic acid, blood sugar) will be performed every day as usual during intensive therapy.

DETAILED DESCRIPTION:
Despite the fact that interventional therapy of vascular lesions (endovascular and hybrid procedures) is becoming more and more common, angioplasties involving major vessels have to be still managed as surgical procedures associated with extreme high demand for transfusion, this applies especially to acute rupture of aortic aneurysm, aortic dissection, aortobifemoral bypass and certain elective procedures where conventional open surgery is the only therapeutic option. Due the generalised atherosclerosis typical for most vascular surgical patients as well as the vulnerability of vessel wall, major blood loss has to be taken in account even during elective surgeries with minimally invasive techniques. In the event that excessive bleeding would occur, conversion to open surgery may be necessary, for this reason the preparation and perioperative care of patients undergoing interventional surgery have to be performed in the same manner as its is prescribed for open aorta operations.

The bleeding risk associated with the above surgical procedures is increased by the fact that the majority of patients affected are on a single or in some cases on double antiplatelet therapy, and/or receive prolonged anticoagulation treatment. Discontinuation of the treatments is expensive and, in case of indication for acute surgery, may not always be carried out.

Previous bleeding history, current drug therapy, evaluation of coagulation status (prothrombin time, activated partial thromboplastin time, thrombin time, fibrinogen) and blood count screening using conventional laboratory tests are part of preoperative preparations. Control of platelet function is always indicated in case of positive anamnesis (inherited or acquired thrombocytopathy, anamnestic information on bleeding complication, skin symptoms suggesting haemophilia), but is not performed routinely. Preoperative normalization of possible abnormalities as well as optimalization of drugs affecting haemostasis, so the reduction of bleeding risk to the minimum are of essential importance, however, we do not always have enough time for it. In cardiovascular surgery, withdrawal of aspirin and/or clopidogrel therapy increases the risk of thrombosis; continuation of aspirin and/or clopidogrel therapy increases the risk of bleeding. In our own practice, in case of elective vascular surgical procedures, aspirin therapy will be continued, but clopidogrel will be stopped 5-7 days prior to surgery, according to the European recommendations. When a patient with prolonged anticoagulant therapy is at high risk for embolism, his medication will be switched to low molecular weight heparin. In case the surgery is performed under ongoing antiplatelet therapy, transfusion of thrombocyte concentrate may also be necessary.

In the European guidelines, the application of transfusion algorithms and protocols incorporating predefined intervention triggers to guide haemostatic intervention during preoperative bleeding are recommended, as well as viscoelastic point-of-care tests (POCT). In lack of the latter, the Hungarian recommendation suggests the application of conventional monitoring assays, however, they give an poor assessment picture with associated with significant time delay, therefore have to be considered inadequate in case of excessive bleeding.

At first, it has to be definitely cleared whether the blood loss is caused by haemostatic or surgical source. In the meantime, however, maintenance of normothermia, prevention of acidosis and normalisation of ionized calcium level are of significant importance. In case of active bleeding the targeted value of systolic blood pressure is 80-100 mmHg, that of haemoglobin concentration 7-9 g/dl. The restrictive transfusion strategy is aimed at decreasing the number of allogeneic transfusions which are regarded as a form of tissue transplantation to the possible minimum.

The first step for optimal restoration of the function of haemostasis system has to be the regulation of the concentration of fibrinogen in the blood plasma, using either conventional laboratory tests or point-of-care testing. Fibrinogen is synthesized in the liver and will not be stored; it has the highest concentration among all coagulation factors (3 g/l). During blood loss, its concentration decreases and reaches the crucial level (<2 g/l) most rapidly. It is essential that besides erythrocyte (RBC) concentrate fresh frozen plasma (FFP) has also to be given (RBC:FFP=2:1) in a timely manner, in a fixed proportion. In case of excessive blood loss and transfusion, administration of thrombocyte concentrate is also necessary.

Aim of the study Comparative study on efficacy of haemostatic therapy guided either by standard laboratory parameters or point-of-care testing in patients undergoing vascular surgical procedures.

Study design Prospective randomised clinical trial

Patients Inclusion criteria Patients scheduled for elective and acute open aorta surgery or undergoing acute aorta surgery with minimally invasive techniques and were provided treatment in the operating theatre and/or ICU attached to perioperative care, they must be at least 18 years of age and written informed consent was obtained from the patient or his/her legal representative.

Randomisation technique:

Patients will be randomly assigned to each of two treatment groups using sealed envelopes:

* Patient group 1: haemostasis strategy guided by conventional coagulation tests.
* Patient group 2: transfusion algorithm guided by viscoelastic POC tests and algorithms.

Exclusion criteria:

* patients under 18 years of age
* informed consent not provided
* congenital coagulation factor deficiency
* congenital thrombocytopathy

Discontinuation criteria:

* death of patient
* withdrawal of consent by the patient or his/her relative

Assessment of parameters Conventional coagulation laboratory tests In the preanalytical phase consisting of steps within and outside the laboratory we have to face a great number of influence factors which can be of critical importance concerning the result of the lab test (e.g. quality of blood sampling tube, method of sampling, appropriate amount of sample, haemolysis, lipaemia). The time-consuming nature of these tests may cause problems primarily in case of massive bleeding. It is not the same blood that circulates in the patient's organism by the time we receive the result. Another disadvantage is that only a few steps of coagulation cascade are investigated. The tests are performed using the plasma separated by centrifugation of blood. Information regarding reactions on the surface of activated platelets, fibrin polymerisation, clot firmness and fibrinolysis cannot be obtained.

Routinely monitored parameters:

* Prothrombin time (PT)/ International normalized ratio (INR): extrinsic coagulation pathway and final common pathway.
* Activated partial thromboplastin time (aPTT): intrinsic coagulation pathway and final common pathway.
* Thrombin Time (TI): reflects the speed of conversion of fibrinogen to fibrin.
* Fibrinogen: amount of fibrinogen in the blood plasma.
* Blood count (platelet number ) Point-of-care methods Point-of-care tests using whole blood provide information within a short time, including the patient's haemostatic status. These benefits are associated with many advantageous features such as small place demand, simply use, no need of maintenance; centrifugation is not required, the reagents are ready to use, some tests can be stored at room temperature.

Viscoelastic tests Viscoelastic tests used for global haemostasis assays are thromboelastography (TEG) and rotational thromboelastometry (ROTEM). The original method has been developed by Harter in 1948 in Heidelberg, initially for analysis of not anticoagulated blood. Viscoelastic tests provide information on primary haemostasis (platelet adhesion and aggregation), thrombin generation, thrombus formation and fibrinolysis, thus, on every steps of haemostasis. Informative analysis in case of patients who are on prolonged heparin therapy can also be accomplished.

Disadvantages of viscoelastic coagulation POC tests include indirectly obtained information on the platelet function, furthermore, the role of endothelium is not recognizes and the characteristics of blood flow are disregarded.

During TEG/ROTEM analysis a pin is dipped into a sample of whole blood - to be given in a cuvette of not physiological surface - and the coagulation becomes activated. Cuvette and sensor move relative to each other. In TEG, the movement is initiated from the cup, in ROTEM the pin is oscillated and the cuvette remains fixed. Increasing viscosity of blood and enhancing stability of clot being formed induce a change of elasticity. This process affects the motion of the sensor that is detected by light reflection changes. The two methods are equivalent and can be considered as mutual alternatives.

The tested parameters provide information on the starting time of clotting process, the clot formation, stabilisation and quality as well as fibrinolysis.

The efficacy of viscoelastic POC tests have been confirmed by several clinical studies, primarily in the field of cardiac surgery, liver transplantation, and traumatology. As per the published data, the number of allogeneic transfusions and postoperative blood loss decreased significantly.

Parameters of ROTEM analysis:

* Clotting time (CT): Time elapsed from beginning of test until the starting time of clotting.
* Clot formation time (CFT): Time to reach 20 mm amplitude from the starting time of clotting.
* Maximum clot firmness (MCF): Provides information on firmness of clot.
* Maximum lysis (ML): Provides information on loss of clot firmness.

Analysis of platelet aggregation Platelet aggregation inhibitors (e.g. aspirin [acetylsalicylic acid], ticlopidine, clopidogrel), significantly decrease the aggregation ability of platelets or may even completely terminate it. During examination, several platelet aggregation agents will be added to the platelet-rich plasma prepared appropriately and the aggregation induced this way will be measured using an impedance aggregometer. The device measures the change of electric resistance between the two electrodes dipped into the blood sample in relation to time.

Most commonly it is applied for adjustment of antiplatelet therapy and monitoring the efficacy of the substance. It is suitable for highly sensitive detection of aspirin, clopidogrel, prasugrel and IIb/IIIa-receptor antagonists.

Now there are literary data also in respect of its efficacy in respect of predicting the probability of coronary stent thrombosis, as well as that of bleeding and the need of transfusion in cardiac surgery. Still, it is not recommended to routinely use this device in the perioperative care of any and all patients. At the same time, however, in case of patients at risk (e.g. positive bleeding anamnesis, treatment with platelet-aggregation inhibiting drugs) it is able to identify and to help diagnose a possible platelet disfunction.

Routinely monitored parameter:

• Area Under the Curve (AUC): Indication of platelet activity. The results calculated by the software are the mean values of data of the several curves.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective and acute open aorta surgery or undergoing acute aorta surgery with minimally invasive techniques and were provided treatment in the operating theatre and/or ICU attached to perioperative care
* they must be at least 18 years of age
* written informed consent was obtained from the patient or his/her legal representative.

Exclusion Criteria:

* patients under 18 years of age
* informed consent not provided
* congenital coagulation factor deficiency
* congenital thrombocytopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The number of blood products used | 24 hours
Amount of perioperative bleeding | 24 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785